CLINICAL TRIAL: NCT00636948
Title: Rectal Cancer Trial On Defunctioning Stoma
Acronym: RECTODES
Status: Completed | Type: Observational
Sponsor: Rectal Cancer Trial on Defunctioning Stoma Study Group (Other)
Responsible Party: Peter Matthiessen, MD, PhD, Department of Surgery, Örebro University Hospital
Other Study IDs: Dnr 99039
Record Dates: First submitted 2008-02-11; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer surgery; Symptomatic anastomotic leakage; Defunctioning stoma; TME surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The hypothesis of the present trial was that the use of a defunctioning loop stoma reduces the rate of symptomatic anastomotic leakage from 15% to 7.5% after low anterior resection of the rectum for cancer.

DETAILED DESCRIPTION:
The assumption that a defunctioning loop stoma reduces symptomatic anastomotic leakage from 15% to 7.5%, with a level of statistical significance of 5% and a statistical power of 80%, requires randomization of 220 patients.

ELIGIBILITY:
Inclusion Criteria:

* Absence of intraoperative adverse events according to the study protocol and the operating surgeon.

Exclusion Criteria:

* Presence of intraoperative adverse events according to the study protocol and the operating surgeon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for rectal cancer in whom low anteriror resection with or without preoperative adjuvant treatment was the planned treatment, who did not have any intraoperative adverse events and who had accepted participation.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 1999-12; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Symptomatic anastomotic leakage following low anterior resection of the rectum for cancer with and without a defunctioning stoma. Anorectal function after one and five years without defunctioning stoma. | 30 days, one year and five years.

SECONDARY OUTCOMES:
Reoperation within 30 days of initial surgery. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rune Sjödahl, MD, PhD, Study Chair — Department of Surgery, Linköping University Hospital
Locations (1):
- Department of Surgery, Linköping University Hospital, Linköping, Sweden

REFERENCES:
- [Result] Matthiessen P, Hallbook O, Rutegard J, Simert G, Sjodahl R. Defunctioning stoma reduces symptomatic anastomotic leakage after low anterior resection of the rectum for cancer: a randomized multicenter trial. Ann Surg. 2007 Aug;246(2):207-14. doi: 10.1097/SLA.0b013e3180603024. PMID 17667498
- [Derived] Floodeen H, Hallbook O, Rutegard J, Sjodahl R, Matthiessen P. Early and late symptomatic anastomotic leakage following low anterior resection of the rectum for cancer: are they different entities? Colorectal Dis. 2013 Mar;15(3):334-40. doi: 10.1111/j.1463-1318.2012.03195.x. PMID 22889325
- [Derived] Matthiessen P, Lindgren R, Hallbook O, Rutegard J, Sjodahl R; Rectal Cancer Trial on Defunctioning Stoma Study Group. Symptomatic anastomotic leakage diagnosed after hospital discharge following low anterior resection for rectal cancer. Colorectal Dis. 2010 Jul;12(7 Online):e82-7. doi: 10.1111/j.1463-1318.2009.01938.x. Epub 2009 Jul 7. PMID 19594606